CLINICAL TRIAL: NCT01634984
Title: The Diagnostic Technology Applied Research of CDK5RAP2 in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CIH-ZHJ-201205001
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: expression of CDK5RAP2
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Selected 400 cases of women with primary breast cancer who were treated with operation randomly, then detect the expression of CDK5RAP2 of cancer tissue. At the same time randomly selected 100 women with primary breast cancer who were under neoadjuvant chemotherapy. Detect the expression of CDK5RAP2 before and after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The investigators selected 400 cases of women with primary breast cancer who were treated with operation randomly,then detect the expression of CDK5RAP2 of cancer tissue. At the same time randomly selected 100 women with primary breast cancer who were under neoadjuvant chemotherapy. Detect the expression of CDK5RAP2 before and after neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Pathological confirmation of breast cancer
3. Tumor stage(TNM):T2-4bN0-3M0
4. ER(+) and/or PR(+).
5. Premenopausal woman.
6. Age≥40 years
7. Measurable disease as per RECIST criteria
8. Karnofsky≥70
9. Laboratory criteria:

   * PLT≥100*109/L
   * WBC≥4000/mm3
   * HGB≥10g/dl
   * ALT and AST<2*ULN

Exclusion Criteria:

1. Presence of metastatic disease.
2. Inflammatory breast cancer.
3. Bilateral breast cancer.
4. previous chemotherapy or hormonal therapy for current breast neoplasm.
5. other malignant tumor (concurrent or previous).
6. Pregnant woman.
7. Hypersensitive to any drug in CEF regimen or any ingredient of Zoladex.
8. Any severe systemic disease contraindicating chemotherapy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 500 patients with breast cancer
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhang, Pro., Study Chair — Tianjin Cancer Hospital
Locations (1):
- Jin Zhang, Tianjin, China